CLINICAL TRIAL: NCT00038415
Title: A Phase I/II Trial of Idiotypic Vaccination for Chronic Lymphocytic Leukemia Using a Genetic Approach
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Vaccine unavailable.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM99-412
Record Dates: First submitted 2002-05-30; First posted 2002-05-31 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Leukemia, Lymphocytic, Chronic
Keywords: Chronic Lymphocytic Leukemia; CLL; Binet Stage A; Vaccination; Idiotypic; Genetic; Deoxyribonucleic acid; DNA
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental)
  Interventions: Biological: CLL vaccine using DNA plasmid vector

INTERVENTIONS:
Biological: CLL vaccine using DNA plasmid vector

SUMMARY:
The goal of this clinical research study is learn if a vaccine that contains the patient's own cancer cell immunoglobulin can shrink or slow the growth of Chronic Lymphocytic Leukemia (CLL). This clinical trial is a dose escalation study in which the safety of this vaccine will be studied. This is a dose escalation study in which each patient will receive vaccine at one dose level. Patients will be injected with a fragment of Deoxyribonucleic acid (DNA) containing the sequence of their own immunoglobulin gene. Patients will be required to have their diagnosis of CLL and stage confirmed prior to initiating vaccination. After vaccination patients will receive clinical and immunologic evaluation, including both humoral and cellular responses. The investigator will be assessing the patient's immune response or whether the patient's body recognizes the DNA vaccine. In addition, side effects and reactions to the vaccine will be evaluated.

DETAILED DESCRIPTION:
OBJECTIVES:

1. To determine if patients with Binet Stage A CLL generate an immune response to an antigen delivered by a DNA vaccine.
2. To determine if patients with Binet Stage A CLL generate an immune response to a tumor derived antigen delivered by a DNA vaccine.
3. To determine the optimal dose of DNA vaccine to obtain anti-idiotype immune responses.
4. To characterize any adverse effects of idiotypic vaccination with a DNA vaccine.
5. To determine if DNA idiotypic vaccination is capable of inducing remission in Binet´s Stage A CLL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Binet Stage A Chronic Lymphocytic Leukemia (CLL)
* WHO performance status of 2 or less.
* A life expectancy of at least one year.
* Greater than 18 years of age.
* Availability of CLL cells which can be used for DNA extraction and processing.
* A platelet count greater than 100 x 109/l.
* Ability to provide full informed consent.

Exclusion Criteria:

* Previous chemotherapy or radiotherapy.
* Presence of a monoclonal band on serum electrophoresis.
* Presence of clinically significant levels of anti-DNA antibodies, anti-muscle antibodies or rheumatoid factors or who have active autoimmune disease.
* Presence of antibodies to human immunodeficiency virus (HIV) and known carriers of hepatitis B or hepatitis C virus.
* Presence of other serious medical condition e.g. congestive heart failure.
* Presence of other malignancies.
* Pregnancy, lactation, or not using contraceptive measures.
* Concurrent use of other anti-cancer therapy.
* Patients allergic to tetanus vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2001-12; Primary Completion 2004-07 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Continuous reassessment up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Keating, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org